CLINICAL TRIAL: NCT05696548
Title: Phase 2 Study of Nivolumab Plus Lenvatinib for Patients With Unresectable Anaplastic Thyroid Cancer (NAVIGATION Study)
Brief Title: Nivolumab Plus Lenvatinib Against Anaplastic Thyroid Cancer (NAVIGATION)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center Hospital East (Other)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Principal Investigator, Makoto Tahara, Chief, Department of Head and Neck Medical Oncology, National Cancer Center Hospital East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YCU18001; JapicCTI-194835 (Registry Identifier: JAPIC Clinical Trials Information)
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Anaplastic Thyroid Cancer
Keywords: Nivolumab; Lenvatinib; Anaplastic Thyroid Cancer
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — lenvatinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lenvatinib plus Nivolumab (Experimental): Step 1: 3 patients, Step 2: 48 patients
  Interventions: Drug: Lenvatinib; Drug: Nivolumab

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib will be administered at a dose of 24mg as oral dose, one a day
Drug: Nivolumab — Nivolumab will be administered at a dose of 240mg as a 30-minutes IV infusion, every 2 weeks

SUMMARY:
This study is an open-label phase 2 study to evaluate the safety and efficacy of Nivolumab plus Lenvatinib in patients with unresectable anaplastic thyroid cancer.

DETAILED DESCRIPTION:
This study is an open-label phase 2 study to evaluate the safety and efficacy of Nivolumab plus Lenvatinib in patients with unresectable anaplastic thyroid cancer according to the following steps.

Step 1 will evaluate the dose-limiting toxicities (DLT) of Nivolumab plus Lenvatinib in patients with unresectable anaplastic thyroid cancer.

Step 2 will evaluate the safety and efficacy of Nivolumab plus Lenvatinib in patients with unresectable anaplastic thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed as anaplastic thyroid cancer
2. Unresectable anaplastic thyroid cancer
3. Have measurable lesions defined by the RECIST version 1.1
4. Have adequate organ function
5. Cardiac function test within 28 days before enrollment 12-lead electrocardiogram no clinically significant abnormality as shown below: heart disease, severe arrhythmia, etc.
6. Patients who are 20 years or older
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
8. Ability to swallow oral medications
9. Women of childbearing potential
10. Life expectancy of more than 90 days
11. Have signed written informed consent to participate in this study

Exclusion Criteria:

1. Active brain metastases or leptomeningeal metastases
2. Diverticulitis or Symptomatic ulcerative disease
3. Treatment required complication of systemic infectious disease
4. Medical history of active, known, or suspected autoimmune disease
5. Complication of pulmonary fibrosis or interstitial pneumonitis
6. Medical history of clinically significant cardiovascular disease within 180 days of initial dose as New York Heart Association (NYHA) class above 2 leveled congestive heart failure, unstable angina, cardiac infarction or cardiac arrhythmia with paroxysmal or required treatment
7. Regardless of usage of antihypertensive drug, systolic blood pressure <=140 mm Hg and diastolic blood pressure <=90 mm Hg
8. Have active double cancer
9. Currently receiving other interventional clinical study treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Step 1: Proportion of subjects with Dose-Limiting Toxicities (DLT) | up to 28 days
  Proportion of subjects with DLT will be defined as the proportion of patients who developed DLT
Step 2: Objective Response Rate (ORR) | Up to 12 months
  ORR will be defined as the proportion of patients achieving complete response (CR) and partial response (PR) as determined according to RECIST ver1.1 by a central review

SECONDARY OUTCOMES:
Proportion of adverse events | Up to 12 months
  For adverse events due to protocol treatment, determine the frequency of worst grades in all courses according to CTCAE v5.0
Overall Survival (OS) | Up to 12 months
  The period will be from the day of enrollment, as the starting date of the computation, to the day of death of any cause.
Progression-Free Survival (PFS) | Up to 12 months
  The registration date is the starting date, and is defined as the period until the progressive disease (PD) or death of any cause occurs.
Best Overall Response (BOR) | Up to 12 months
  BOR is the best response recorded from the start of the study treatment until the end of treatment
Disease Control Rate (DCR) | Up to 12 months
  DCR will be defined as the proportion of patients achieving CR, PR or stable disease (SD).
Clinical Benefit Rate (CBR) | Up to 12 months
  DCR will be defined as the proportion of patients achieving CR, PR or SD lasting at least 11 months.
Quality of life by EuroQol 5 dimensions 5-level (EQ-5D-5L) | Up to 12 months
  Quality of life will be evaluated by EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Tahara, MD, PhD, Study Director — National Cancer Center Hospital East; Iwao Sugitani, MD, PhD, Study Chair — Nippon Medical School Hospital; Naomi Kiyota, MD, PhD, Study Chair — Kobe University Hospital
Locations (10):
- Japan (10):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hokkaido University Hospital, Hokkaido, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - National Cancer Center Hospital, Tokyo, Tokyo
  - Nippon Medical School Hospital, Tokyo, Tokyo

IPD SHARING:
Plan to Share IPD: No